CLINICAL TRIAL: NCT05221658
Title: An Open-label, Multicenter , Phase II Clinical Study to Evaluate the Efficacy and Safety of HLX07 ( Recombinant Humanized Anti-EGFR Monoclonal Antibody Injection) Combination Therapy or Monotherapy in Patients With Locally Advanced, Unresectable or Metastatic Esophageal Squamous Cell Carcinoma (ESCC)
Brief Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of HLX07 Combination Therapy or Monotherapy in Patients With Advanced ESCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX07-ESCC201
Record Dates: First submitted 2022-01-22; First posted 2022-02-03 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: ESCC or Esophageal Adenosquamous Carcinoma
MeSH Terms: interventions — HLX07

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): As first-line therapy
  Interventions: Drug: HLX07+HLX10+ Cisplatin+5-FU
- Arm B1 (Experimental): EGFR H score ≥ 200, as third-line or above therapy
  Interventions: Drug: HLX07
- Arm B2 (Experimental): EGFR H score <200, as third-line or above therapy
  Interventions: Drug: HLX07

INTERVENTIONS:
Drug: HLX07+HLX10+ Cisplatin+5-FU — HLX07 1000mg + HLX10 200mg + Cisplatin 50 mg/m2 + 5-FU 2400mg/m2
  Arms: Arm A
Drug: HLX07 — HLX07 1000mg iv Q2w
  Arms: Arm B1; Arm B2

SUMMARY:
This study is conducted in patients with Locally advanced, unresectable, or metastatic esophageal squamous cell carcinoma (ESCC) or esophageal adenosquamous carcinoma. This study includes three arms: A, B1, and B2. Arm A will receive HLX07 combination therapy with HLX10 and Chemotherapy (Cisplatin+5-FU) as first line treatment. Arm B (Patients with EGFR expression H score ≥ 200) and Arm C (Patients with EGFR expression H score < 200) will receive HLX07 monotherapy as third-line or above treatment. All of eligible patients will receive study drug treatment until loss of clinical benefit, unacceptable toxicity, death, withdrawal of informed consent (whichever occurs first, HLX10 treatment up to 2 years).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all of the following criteria are allowed to be enrolled into this study:

  * Volunteer to participate in this clinical study; completely understand and know this study as well as sign the informed consent form (ICF); be willing to follow and be able to complete all study procedures;
  * Age ≥ 18 years and ≤ 75 years when ICF is signed;
  * Histopathologically or cytologically confirmed diagnosis of locally advanced, unresectable or metastatic esophageal squamous cell carcinoma (ESCC) or esophageal adenosquamous carcinoma.
  * Subjects in Arm B1 and Arm B2 must provide eligible tumor tissue for EGFR expression level determination： Arm B1: Subjects with EGFR expression H score ≥ 200 confirmed by central laboratory immunohistochemistry (IHC) in tumor tissue.

Arm B2: Subjects with EGFR expression H score < 200 confirmed by central laboratory IHC.

* prior therapy: Arm A: Never received systemic anti-tumor drug therapy before. Exception: for patients who have received neoadjuvant/adjuvant treatment, the time from the last treatment to recurrence or progression can be screened for more than 6 months; Arms B1 and B2: Failed or intolerant to prior systemic anti-tumor therapy (at least 2 lines).
* According to the curative effect evaluation criteria in solid tumors (RECIST) v1.1, assessed by the investigator with at least one measurable lesions (such as esophageal cavity structure not as measurable lesions), measurable lesions should be not received radiotherapy, etc (lesions located in the usual radiation area, if confirm progress, can also be selected as the target lesion);
* Within 7 days before the first use of the study drug, ECOG: 0 ~ 1;
* Expected survival 12 weeks;
* The functions of the vital organs meet the following requirements (no blood transfusion, cytokine growth factor, or platelet raising drugs are allowed within 14 days before the first use of the study drugs); Absolute neutrophil count (ANC) ≥1.5×109/L platelet≥ 100×109/L; Hemoglobin≥ 90g/L; Serum albumin≥ 30g/L; Total bilirubin≤ 1.5 ULN, ALT, AST and/or ALP≤ 2.5 ULN;ALT and/or AST≤ 5 ULN in the presence of liver metastasis;If there is liver metastasis or bone metastasis ALP≤ 5 ULN; Serum creatinine ≤1.5 ULN or creatinine clearance > 50 mL/min (Cockcroft-Gault formula); APTT, INR and PT ≤1.5 ULN;
* For fertile female subjects, the serum pregnancy test must be negative within 7 days before the first dose.
* With fertile women subjects, and the partner for childbearing age women of male subjects, needs during the therapy, and after the last use HLX10 / placebo at least 6 months and the last time to use at least 6 months after chemotherapy using an approved by the medical contraception (such as intrauterine device, the pill or condoms)

Exclusion Criteria:

* Subjects who meet any of the following criteria are not allowed to be enrolled in this study:

  * A history of gastrointestinal perforation and/or fistula within 6 months prior to the first administration;
  * Obvious invasion of tumor into adjacent organs (aorta or trachea) of esophageal lesions leads to high risk of bleeding or fistula;3. Subjects after endotracheal stent implantation;
  * Uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage;
  * Previous allergies to monoclonal antibody, HLX10, 5-fu, cisplatin and other platinum drugs;
  * Have received any of the following treatments:

A.Prior systemic anti-EGFR monoclonal antibody therapy Previous treatment with anti-pd-1 or anti-pd-L1 antibodies （Arm A）; B. Have received any research drugs within 4 weeks before the first use of the study drugs; C. Be enrolled in another clinical study at the same time, unless it is an observational (non-interventional) clinical study or a follow-up interventional clinical study; D. Receive the final anticancer treatment within 4 weeks before the first use of the study drug;Palliative radiotherapy for bone metastases was allowed and was completed 2 weeks before the first dose.Radiotherapy covering more than 30% of the bone marrow area is not allowed within 28 days before the first dose.

E. Subjects who require systemic treatment with corticosteroids (> 10 mg/ day prednisone therapeutic dose) or other immunosuppressive agents within 14 days prior to the first use of the study drug;In the absence of active autoimmune disease, inhalation or topical use of steroids is permitted, and the therapeutic dose of prednisone 10mg/ day is allowed.

F. Those who have received the anti-tumor vaccine or the live vaccine within 4 weeks before the first dose of the study drug; G. Have undergone major surgery within 28 days prior to the first use of the study drug. Major surgery in this study is defined as requiring at least 3 weeks of postoperative recovery time before being able to receive the surgery treated in this study.Tumor puncture or lymph node biopsy were allowed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 2 years
  Objective response rate by IRRC/INV assessment per RECIST
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 2 years
  Progression-free survival by IRRC/INV assessment per RECIST

SECONDARY OUTCOMES:
OS | from the date of first dose unitl the date of death from any cause，assessed up to 2 years
  Ooverall survival
DOR | from the date when CR or PR (whichever recorded earlier) is firstly achieved until the date when disease progression or death is firstly recorded (whichever occurs earlier),assessed up to 2 years
  Duration of response

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Cancer Hospital Chinese Academic of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Cancer Hospital Chinese Academic of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong
  - Anyang Cancer Hospital, Anyang, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - Henan Cancer Hospital & Affiliated Cancer Hospital of Zhengzhou University, Zhenzhou, Henan
  - Hunan Cancer Hospitla, Changsha, Hunan
  - Jiangsu Cancer Hospital & Jiangsu Institute of Cancer Research, Nanjing Medical University Affiliated Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu People Hospital & The First Affiliated with Nanjing Medical University, Nanjing, Jiangsu
  - Xuzhou Center Hospital, Xuzhou, Jiangsu
  - Shandong Cancer Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Yunnan Cancer Hospital & The Third Affiliated Hospital of Kunming Medical University & Yunnan Cancer Center, Kunming, Yunnan

REFERENCES:
- [Derived] Liu Y, Wang Y, Zhu Y, Wu T, Liu Z, Zhou J, Yuan Y, Yang M, Liu B, Tan Z, Zhuang W, Chen J, Li N, Wang Y, Hu X, Wang L, Yu H, Wang Q, Zhu J, Huang J. HLX07 alone or combined with serplulimab, cisplatin and 5-fluorouracil for advanced esophageal squamous cell carcinoma: A phase 2 study. Cancer Commun (Lond). 2024 Dec;44(12):1431-1443. doi: 10.1002/cac2.12621. Epub 2024 Oct 24. PMID 39446605